CLINICAL TRIAL: NCT04775251
Title: Effect of Scapular Upward Rotation Exercises on Neural Tissue Mechanosensitivity in Subjects With Deperessed Scapular Alignment
Brief Title: Scapular Upward Rotation Exercises for Subjects With Deperessed Scapular Alignment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doha Hamed Moustafa Al-Afifi, Principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/002640
Record Dates: First submitted 2021-02-06; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Scapular Dyskinesis
Keywords: Neural tissue mechanosensitivity; Depressed Scapular Alignment; Scapular upward rotation exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one group (Experimental): The treatment program consisted of upward rotation exercises for 3 sessions/week, for 6 weeks.
  Interventions: Other: Upward rotation exercise

INTERVENTIONS:
Other: Upward rotation exercise — Treatment for correction of depressed scapular Alignment by exercise ( Upward Rotation Exercises) for 6 weeks.

SUMMARY:
It was hypothesized that:

There is no statistical significant effects of a scapular vupward rotation exercise (SURE) on scapular alignment in subjects with scapular downward rotation syndrome (SDRS).

There is no statistical significant effects a scapular upward rotation exercise (SURE) on mechanosensitivity of the upper limb peripheral nervous system in a depressed scapular alignment subjects.

There is no statistical significant effects a scapular upward rotation exercise (SURE) on pressure Pain Threshold in a depressed scapular alignment subjects.

There is no statistical significant effects a scapular upward rotation exercise (SURE)on Strenght Duration Curve measurement in a depressed scapular alignment subjects.

DETAILED DESCRIPTION:
This study was conducted to investigate the effects of scapular upward rotation exercises on strength duration curve and pressure pain threshold (PPT) in subjects with scapular downward rotation syndrome.

Thirty subjects with age range of 18 to 30 years with scapular downward rotation were recruited in this study.

Thirty subjects of both gender with scapular downward rotation were recruited in this study.

All recruited subjects were examined to exclude defined pathological conditions.

All subjects were assessed by screening examination for downward rotation of scapula.

Pressure pain threshold was measured using pressure algometer. Mechanosensitivity of neural tissue was measured using neurodynamic test. Pain was measured using strength-duration (SD) curve. Treatment program consisted of 3 sessions/week, for 6 weeks. All measurements were taken pre and post the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* University population were screened for subjects with scapular downward rotation, those who met the following criteria was recruited in this study. The inclusion criteria for subject selection in this study was based on the literature (Caldwell et al., 2007; Ha et al., 2011) which included:

  1. The scapula was downwardly rotated by visual appraisal.We examined the root of spine of scapulae (superior angle) and inferior angle of scapulae. If scapulae was downwardly rotated, inferior angle closer to spine than root of spine of scapulae (superior angle).
  2. The clavicle appeared to be horizontal or the acromioclavicular joint was lower than the sternoclavicular joint by visual appraisal.
  3. The vertebral borders of the scapula was less than 3 inches from the spine by tape measure.

Exclusion Criteria:

* Subject who has any of the following criteria was excluded from the study:

  1. Subjects with cervical spinal fractures.
  2. Neck-rotation ROM of <20º.
  3. Radiating pain to an upper extremity.
  4. Scoliosis.
  5. Leg length discrepancy.
  6. A history of unresolved cancer.
  7. Diabetes Miletus.
  8. Polyneuropathy.
  9. Myofascial Pain Syndrome.
  10. Fibromyalgia.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-28 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Neural excitability | Strenght-duration curve for neural excitability is measured before starting the treatment.Strenght-duration is measured after application of 6 weeks treatment program.
  Neural excitability measured by Strenght-duration cruve.

SECONDARY OUTCOMES:
Pressure pain threshold | All measurements were taken pre and post the treatment period (6 weeks).
  Pressure pain threshold was measured using pressure algometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ragiaa Kamel, Study Chair — Basic Science Department, Faculty of Physical Therapy, Cairo University; Amr Shalaby, Study Director — Basic Science Department, Faculty of Physical Therapy, Cairo University

IPD SHARING:
Plan to Share IPD: Yes
I commit to share the results of this study within 3-6 months of publicatin.
Time Frame: I commit to share the results of this study within 3-6 months of publication.